CLINICAL TRIAL: NCT04086537
Title: Association Between BMPR2 Mutations and Iron Metabolism in Pulmonary Arterial Hypertension Patients: an Explorative Cross-sectional Study
Brief Title: BMPR2 Mutations and Iron Metabolism in Pulmonary Arterial Hypertension
Acronym: AMIA
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: University Hospital Heidelberg (Other); Hannover Medical School (Other); University Hospital Carl Gustav Carus (Other); University of Leipzig (Other); University of Giessen (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med., Heidelberg University
Other Study IDs: 2019-03IM
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; BMPR2; Iron Metabolism; Hepcidin; Mutations
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Routine clinical laboratory investigations: Iron metabolism:Hepcidin, iron, ferritin, interleukin 6, transferrin, circulating soluble transferrin receptor levels; Hematology:Leucocytes, erythrocytes, hemoglobin, hematocrit, platelets; Substrates: Bilirubin, cholesterol, triglycerides, creatinine, uric acid, urea, total protein, albumin, glucose; Electrolytes:Sodium, potassium, calcium, chloride; Enzymes:serum glutamate oxaloacetate transaminase (SGOT), serum glutamate pyruvate transaminase (SGPT), Gamma-GT, Glutamate Dehydrogenase (GLDH), alkaline phosphatase (AP), lactate dehydrogenase (LDH), creatine kinase (CK); Others:international normalized Ratio (INR), partial thromboplastin time (PTT); Biomarkers:C-reactive Protein (CRP), NT-proBNP; BMPR2 expression with real time quantitative polymerase chain reaction (qPCR), RNA extraction with Quiacube, cDNA production using Transcriptor First Strand cDNA Synthesis Kit; Laboratory assessments will be determined locally on-site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BMPR2-mutation carriers: Patients affected by pulmonary arterial hypertension (PAH) with already determined BMPR2 mutation status (hereditary PAH, HPAH) or patients with idiopathic PAH (IPAH) and other forms of PAH who are newly diagnosed within the duration of the study and resulted positive for mutation at the routinely-performed (according to current guidelines) BMPR2 analysis.
  Interventions: Diagnostic Test: hepcidin levels and BMPR2 expression
- non-BMPR2 mutation carriers: Patients affected by Pulmonary arterial hypertension (PAH) who resulted negative at the routinely-performed (according to current guidelines) BMPR2 analysis (Idiopathic PAH, IPAH) or patients with Idiopathic PAH (IPAH) and other forms of PAH who are newly diagnosed within the duration of the study and resulted negative for mutation at the routinely-performed (according to current guidelines) BMPR2 analysis.
  Interventions: Diagnostic Test: hepcidin levels and BMPR2 expression
- healthy controls: Healthy controls free of heart and lung disease or any comorbidities affecting iron metabolism. This control group will be age and gender matched to non-BMPR2 mutation carriers.
  Interventions: Diagnostic Test: hepcidin levels and BMPR2 expression

INTERVENTIONS:
Diagnostic Test: hepcidin levels and BMPR2 expression — Samples will be collected in the three groups. Hepcidin levels will be measured in serum using ELISA and BMPR2 expression will be assessed as previously described using real time-qPCR

SUMMARY:
Previously characterised PAH patients, including idiopathic, heritable and other forms of group 1 PAH with and without BMPR2 mutation which have already been analysed and are regularly seen in the Center for Pulmonary Hypertension may be contacted to participate in the study. Clinical and laboratory values will be collected prospectively.

Patients with IPAH/HPAH and other forms of PAH who are newly diagnosed within the duration of the trial will receive routine diagnostic workup including the routine information about a possible BMPR2 mutation analysis for IPAH/HPAH patients according to guidelines.

During their routine visit the patients' medical history will be obtained and physical examination will be conducted. Moreover, an electrocardiogram (ECG), determination of World Health Organization (WHO)-functional class, laboratory testing (NT-proBNP and routine laboratory), echocardiography will be routinely carried out. BMPR2 expression levels will be measured in blood samples. Additionally, laboratory samples will be collected for analysis of further parameters reflecting iron metabolism such as hepcidin, ferritin, iron levels, IL6 and circulating soluble transferrin receptor Levels.

In addition, healthy controls will be invited to participate in this study to obtain comparable levels of hepcidin and BMPR2 pathway members.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a rare disease characterized by an increase in pulmonary arterial pressure and pulmonary vascular resistance, which result in right heart hypertrophy and decompensation. It crucially affects exercise capacity, quality of life and prognosis. Idiopathic and heritable forms of PAH (IPAH and HPAH) are often associated with mutations of the bone morphogenetic protein receptor 2 (BMPR2) accompanied by disease development at an earlier age, more severe hemodynamic phenotype and a higher mortality rate. Other forms of PAH also show reduced expression levels of BMPR2, even if no BMPR2 mutation has been identified in these patients. Moreover, the balance of iron metabolism was shown to be disturbed in IPAH patients. IPAH patients suffered from iron deficiency with low levels of serum iron concentrations and while at the same time displaying high levels of the iron uptake regulating hormon hepcidin. The hormone hepcidin, which inhibits iron absorption from the intestine, is upregulated by the BMPR2 signaling pathway (via BMP6). The impact of BMPR2 expression on iron homeostasis, however, has not been investigated yet.

Mutation and non-mutation carriers with invasively diagnosed PAH by right heart catheter and under optimized medical therapy will be enrolled in this study. An explicit exclusion criterion is intravenous iron supplementation in the last 2 months to capture their natural iron metabolic status. Subjects will be recruited at the Center for Pulmonary Hypertension at Thoraxklinik Heidelberg University Hospital. The measurement of BMPR2 expression will be performed with real-time polymerase chain reaction. In addition, routine laboratory parameters of iron metabolism and clinical parameters will be statistically correlated with the BMPR2 expression of BMPR2 mutation carriers and non-mutation carriers. Clinical examinations will comprise of routine diagnostic workup. No study specific clinical assessments will be performed. For diagnostic workup, an extended blood analysis for BMPR2 expression will be performed, which is mentioned in the informed consent document.

In addition, healthy controls will be invited to participate in this study.Healthy controls will only receive a blood collection to obtain control values for hepcidin, BMPR2 expression rate and levels of BMPR2 pathway members such as Bone Morphogenetic Protein 2 and 6 (BMP2 and BMP6). They will not receive any further examinations. BMPR2 mutation status will not be investigated. The control group will be age and gender matched to non-BMPR2 mutation carriers.

Therefore, this study aims to investigate whether PAH patients with a reduced expression rate of BMPR2 have altered serum levels of hepcidin and further iron related metabolites compared to PAH patients with normal expression levels and whether these patients present with more pronounced limitations in clinical parameters. This study could help to understand iron metabolism in PAH and generate new therapeutic targets for the treatment of the disease.

ELIGIBILITY:
Inclusion Criteria Patients:

1. Informed consent
2. Male or female PAH, including idiopathic, heritable and other forms of group 1 PAH (according to Nice classification) patients 18-80 years of age
3. Invasively diagnosed PAH by right heart catheter (invasively confirmed diagnosis according to the current PAH definition of valid guidelines at time of initial diagnosis)
4. Optimized medical therapy for PAH (such as endothelin-receptor-antagonists, inhaled prostanoids, phosphodiesterase-5-inhibitors, diuretics and if useful, supplemental oxygen) for at least 2 months before entering the study
5. Able to understand and willing to sign the Informed Consent Form

Inclusion Criteria Healthy Controls:

1. Informed consent
2. Male or female healthy controls 18-80 years of age
3. Able to understand and willing to sign the Informed Consent Form

Exclusion Criteria Patients:

1. Pregnancy or lactation
2. Change in disease-specific medication within 8 weeks before enrolment
3. Intravenous iron supplementation within the preceding 2 months
4. Acute infection
5. Comorbidities affecting iron metabolism such as hemolytic anemias, genetic disorders of hemoglobin, diabetes, systemic cardiovascular disease, sickle cell disease, thalassemia

Exclusion Criteria Healthy Controls:

1. Pregnancy or lactation
2. Intravenous iron supplementation within the preceding 2 months
3. Acute infection
4. Heart or lung disease
5. Comorbidities affecting iron metabolism such as hemolytic anemias, genetic disorders of hemoglobin, diabetes, systemic cardiovascular disease, sickle cell disease, thalassemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: BMPR2-mutation carriers and non-BMPR2 mutation carriers will be asked for participation in the study.
  Healthy controls will be invited to participate in this study to obtain comparable levels of hepcidin and BMPR2 pathway members. This control group will be age and gender matched to non-BMPR2 mutation carriers. They will not receive any further examinations. BMPR2 mutation status will not be investigated.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
The relationship between absolute values of hepcidin levels and BMPR2 expression | at enrollment
  assessed as correlation between BMPR2 expression levels and hepcidin levels
The relationship between hepcidin levels and BMPR2 expression | at enrollment
  analysis of differences of hepcidin levels in BMPR2 mutation carriers and non-carriers (BMPR2 mutation carriers are assumed to have a lower expression level of BMPR2)

SECONDARY OUTCOMES:
Correlation of BMPR2 expression levels with ferritin levels | at enrollment
  Ferritin levels
Correlation of BMPR2 expression levels with transferrin levels | at enrollment
  Transferrin levels
Correlation of BMPR2 expression levels with soluble transferrin receptor saturation and concentration | at enrollment
  Soluble transferrin receptor saturation and concentration
Correlation of BMPR2 expression levels with iron levels | at enrollment
  Iron levels
Correlation of BMPR2 expression levels with red blood distribution cell width | at enrollment
  Red blood distribution cell width
Correlation of BMPR2 expression levels with erythroferrone levels | at enrollment
  Erythroferrone levels
Correlation of BMPR2 expression levels with hemoglobin levels | at enrollment
  Hemoglobin levels
Correlation of BMPR2 expression levels with hematocrit | at enrollment
  Hematocrit
Correlation of BMPR2 expression levels with erythropoietin (EPO) levels | at enrollment
  Erythropoietin (EPO) levels
Correlation of BMPR2 expression levels with C-reactive protein levels | at enrollment
  C-reactive protein levels
Correlation of BMPR2 expression levels with interleukin 6 (IL6) levels | at enrollment
  Interleukin 6 (IL6) levels to approximate inflammation
Correlation of BMPR2 expression levels with NT-proBNP levels | at enrollment
  NT-proBNP levels
Correlation of BMPR2 expression levels with BMP2 messenger ribonucleid acid (mRNA) expression levels | at enrollment
  BMP2 mRNA expression levels
Correlation of BMPR2 expression levels with BMP6 messenger ribonucleid acid (mRNA) expression levels | at enrollment
  BMP6 mRNA expression levels
Correlation of BMPR2 expression levels with overall transcriptomic analysis in blood samples and formalin fixed human PAH lung tissue samples | at enrollment
  overall transcriptomic analysis in blood samples and formalin fixed human PAH lung tissue samples
Correlation of BMPR2 expression levels with BMPR2 protein levels | at enrollment
  BMPR2 protein levels
Correlation of BMPR2 expression levels with BMP2 protein levels | at enrollment
  BMP2 protein levels
Correlation of BMPR2 expression levels with BMP6 protein levels | at enrollment
  BMP6 protein levels
Correlation of BMPR2 expression levels with 6-minute walking distance (6-MWD) | at enrollment
  6-minute walking distance (6-MWD)
Correlation of BMPR2 expression levels with BORG Scale of 6-minute walking distance (6-MWD) | at enrollment
  Borg Scale of 6-minute walking distance (6-MWD)
Correlation of BMPR2 expression levels with WHO functional class | at enrollment
  WHO functional class
Correlation of BMPR2 expression levels with forced vital capacity (FVC) | at enrollment
  forced vital capacity (FVC)
Correlation of BMPR2 expression levels with forced expiratory volume in one second (FEV1) | at enrollment
  forced expiratory volume in one second (FEV1)
Correlation of BMPR2 expression levels with forced expiratory flow (FEV) | at enrollment
  forced expiratory flow (FEV)
Correlation of BMPR2 expression levels with total lung capacity (TLC) | at enrollment
  total lung capacity (TLC)
Correlation of BMPR2 expression levels with diffusion-limited carbon monoxide (DLCo) | at enrollment
  diffusion-limited carbon monoxide (DLCo)
Correlation of BMPR2 expression levels with residual volume | at enrollment
  residual volume, normally accounting for about 25% of total lung capacity
Correlation of BMPR2 expression levels with blood gas analysis including partial pressure of oxygen | at enrollment
  partial pressure of oxygen
Correlation of BMPR2 expression levels with blood gas analysis including partial pressure of carbon dioxide | at enrollment
  partial pressure of carbon dioxide
Correlation of BMPR2 expression levels with blood gas analysis including oxygen saturation | at enrollment
  oxygen saturation
Correlation of BMPR2 expression levels with blood gas analysis including supplemental oxygen "yes" or "no" | at enrollment
  supplemental oxygen "yes" or "no"
Correlation of BMPR2 expression levels with cardiac output (CO) | at enrollment
  cardiac output (CO) measured by right heart catheterization
Correlation of BMPR2 expression levels with cardiac index (CI) | at enrollment
  cardiac index (CI) measured by right heart catheterization
Correlation of BMPR2 expression levels with pulmonary capillary wedge pressure (PAWP) | at enrollment
  pulmonary capillary wedge pressure (PAWP) measured by right heart catheterization
Correlation of BMPR2 expression levels with mixed venous oxygen saturation (SvO2) | at enrollment
  mixed venous oxygen saturation (SvO2) measured by right heart catheterization
Correlation of BMPR2 expression levels with right atrium area (RA-area) | at enrollment
  right atrium area (RA-area) determined by echocardiography
Correlation of BMPR2 expression levels with right ventricle area (RV-area) | at enrollment
  right ventricle area (RV-area) determined by echocardiography
Correlation of BMPR2 expression levels with myocardial performance index (Tei) | at enrollment
  myocardial performance index (Tei) determined by echocardiography
Correlation of BMPR2 expression levels with tricuspid annular plane systolic excursion (TAPSE) | at enrollment
  tricuspid annular plane systolic excursion (TAPSE) determined by echocardiography
Correlation of BMPR2 Expression with systolic pulmonary artery pressure | at enrollment
  systolic pulmonary artery pressure determined by echocardiography
Correlation of BMPR2 Expression with right ventricular function | at enrollment
  right ventricular function determined by echocardiography
Correlation of BMPR2 Expression with left ventricular function | at enrollment
  left ventricular function determined by echocardiography
Correlation of BMPR2 Expression with right ventricular pressure | at enrollment
  systolic, diastolic and mean right ventricular pressure measured by right heart catheterization
Correlation of BMPR2 Expression with pulmonary artery pressure | at enrollment
  systolic, diastolic and mean pulmonary artery pressure measured by right heart catheterization
Correlation of BMPR2 Expression with pulmonary vascular resistance | at enrollment
  pulmonary vascular resistance measured by right heart catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Pulmonary Hypertension at the Thoraxklinik, Heidelberg University Hospital, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No